CLINICAL TRIAL: NCT06749613
Title: Digestive Enzyme Formulation Intervention in Irritable Bowel Syndrome Patients Who Previously Clinically Responded to Mediterranean Low FODMAP Diet: A Single-Arm Clinical Trial
Brief Title: Digestive Enzyme Formulation Intervention in IBS Patients Who Previously Clinically Responded to Mediterranean LFD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Arezina Kasti, Senior Dietitian, Attikon Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ΕΒΔ 185/04-03-2024
Record Dates: First submitted 2024-12-10; First posted 2024-12-27 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Irritable Bowel Syndrome
Keywords: low FODMAP Diet; MED-LFD; digestive enzymes
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- digestive enzymes group (Experimental): Patients will be instructed to use a powder formulation according to manufacturer instructions and according to the meals that they consume per day, for 1 month. To reduce the placebo effect, patients will be misinformed that half will take a placebo formulation, randomly.
  Interventions: Dietary Supplement: digestive enzymes

INTERVENTIONS:
Dietary Supplement: digestive enzymes — A jar or single-dose sachets containing the digestive enzymes in the form of powder will be provided to each patient at the study entry. Patients will be instructed to use the powder formulation according to manufacturer instructions and according to the meals that they consume per day, for 1 month. Participants will be asked to return the jar or the single dose sachets with the remaining product to assess compliance either by weighting the jar or by counting the number of single-dose sachets returned. To reduce the placebo effect, patients will be misinformed that half will take a placebo formulation, randomly. Participants will be asked to return the jar or the single-dose sachets with the remaining product to assess compliance either by weighting the jar or by counting the number of single-dose sachets returned.

SUMMARY:
Irritable bowel syndrome (IBS) is a highly prevalent chronic functional gastrointestinal disorder. The cardinal symptoms include abdominal pain, flatulence, bloating, and changes in bowel habits related to stool frequency and consistency, in the absence of detectable structural and biochemical abnormalities1,2. The prevalence is estimated at 5-10% among different ethnicities3. A low FODMAP diet is the most common dietary intervention with clinically proven benefits in symptom management and quality of life improvement of patients with Irritable Bowel Syndrome (IBS)4. Recently, a dietary digestive enzyme formulation (FODZYME©) claims similar efficacy in symptom management based on an ex-vivo study5. The study aims to examine the clinical efficacy of this formulation in managing IBS symptoms in patients who have previously clinically responded to a low FODMAP diet.

DETAILED DESCRIPTION:
IBS patients who participated in a two-arm clinical trial (ClinicalTrials.gov ID: NCT03997708) and responded to the Mediterranean Diet Adjusted Low FODMAP (MED-LFD) Diet will be considered eligible if their symptoms recurred one year after their initial response to the dietary intervention. Among them, patients without any or mild symptoms, defined as IBS severity scoring system (IBS-SSS) ≤ 175, will be excluded. Moreover, subjects who were randomized to the MED-LFD arm in the previous study, but could not adhere to the dietary intervention, will be included too.

A jar containing the digestive enzymes in the form of powder will be provided to each patient at the start of the study. Patients will be instructed to use the powder formulation according to manufacturer instructions for 1 month. To assess compliance, the weight of each jar will be measured both at the initiation and the end of the study. Patients will also be asked on three different days (one day from the weekend), to estimate the average number of meals per day. Due to the limited sample size (54 patients who received the MED-LFD diet in the previous phase will be screened for eligibility), a control group will be omitted. To reduce the placebo effect, patients will be misinformed that half will take a placebo formulation, randomly.

All patients will be thoroughly trained regarding the proper consumption of the powder (exact dose, timing, etc.), through personal training, videos, leaflets, and other type of training materials.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent.
* Commitment to availability throughout the study period.
* Patients who fulfilled the Rome IV criteria for IBS (IBS-D, IBS-M, IBS-U) participated in the two-arm clinical trial (ClinicalTrials.gov ID: NCT03997708) as responders to the Mediterranean Diet Adjusted to Low FODMAP (MED-LFD) (if their symptoms recurred -with IBS-SSS > 175- one year after their initial response to the dietary intervention).
* Subjects randomized to the MED-LFD arm of the previous study who could not adhere to the dietary intervention.

Exclusion Criteria:

* Patients who did not take part in the aforementioned study
* Patients who were randomized in the NICE group
* Patients with IBS-SSS<175.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-10-10 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Changes in IBS-SSS from baseline to follow-up | 1 month
  Changes in IBS-SSS from baseline to follow-up in the group of patients that have responded to MED-LFD in the past. The IBS-SSS questionnaire consists of 5 specific questions6. Each of the five questions (pain severity, pain frequency, abdominal distension severity, bowel movement satisfaction, quality of life) ranges from a minimum score of 0 to a maximum score of 100, using a visual analog scale (VAS), with total scores ranging from 0 to 500.

SECONDARY OUTCOMES:
Changes in the Gastrointestinal Symptom Rating Scale - IBS version (GSRS-IBS). | 1 month
  The GSRS questionnaire is validated in patients with IBS. GSRS-IBS consists of 13 items, designed to assess gastrointestinal symptoms specifically for IBS patients. Each item is rated based on a 7-point Likert scale (1. "No discomfort at all"; 2. "Minor discomfort"; 3. "Mild discomfort"; 4. "Moderate discomfort"; 5. "Moderately severe discomfort"; 6. "Severe discomfort"; 7. "Very severe discomfort"). The questionnaire has a total score and five subscales (pain, bloating, constipation, diarrhea, and satiety), calculated by summing all questions corresponding to each scale and dividing with the number of questions summed in each scale. Both total and subscale scores are ranging from 1 (no discomfort) to 7 (severe discomfort), with higher scores representing increased symptom burden.
Changes in SF-12. | 1 month
  SF-12 is a 12-item questionnaire used to assess generic health outcomes from the patient's perspective, covering two domains of health outcomes: physical functioning and mental health. The items are weighted and summed to provide physical and mental health scores. The two composite scores are computed using the scores on the questions that range from 0 to 100, with higher score indicating better QoL. SF-12 is validated also in the Greek population.
Changes in IBS-Qol. | 1 month
  The IBS-QoL assesses the degree to which IBS interfered with quality of life over the past 30 days10. It is a self-reported quality of life measure, which includes eight domains, such as dysphoria, interference with activity, body image, health worry, food avoidance, social relations, sexual and relationship issues. Each of them is rated based on a 5-point Likert scale (1. "Not at all"; 2." Slightly"; 3. "Moderately"; 4. "Quite a bit" 5. "Extremely/ A great deal").

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - Attikon University General Hospital, Chaïdári, Athens
  - Attikon University General Hospital, Athens